CLINICAL TRIAL: NCT00422786
Title: A Multi-Centre, Open Label, Phase II Study of the Safety, Efficacy and Pharmacokinetic (PK) Profile of CAP-232 Administered Through Continuous Intravenous Infusion in Patients With Metastatic Kidney Cancer
Brief Title: Phase II Study of CAP-232 in Patients With Refractory Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thallion Pharmaceuticals (Industry)
Responsible Party: Didier Reymond, MD / Vice-President Medical and Clinical Affairs, Thallion Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP_CAP001
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Carcinoma, Renal Cell
Keywords: Refractory Clear Cell Renal Cell Carcinoma; Phase II; Thallion; TLN-232; CAP-232; M2PK
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAP-232 (Experimental): Continuous IV infusion over 21 days at 0.48 mg/kg/day followed by a 7-day rest period.
  Interventions: Drug: CAP-232

INTERVENTIONS:
Drug: CAP-232 — Continuous IV infusion over 21 days at 0.48 mg/kg/day followed by a 7-day rest period
  Other Names: TLN-232

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of CAP-232 in the treatment of patients with previously treated (refractory) renal cell carcinoma

DETAILED DESCRIPTION:
This was a multi-center, open label, single arm study. Approximately 40 patients were initially planned to be recruited.

Each patient was to receive a treatment cycle consisting of CAP-232 via continuous IV infusion over 21 days at 0.48 mg/kg/day followed by a 7-day rest period. Treatment cycles to be repeated in the absence of disease progression or unacceptable toxicity.

Quality of Life questionnaires were to be administered at baseline, after each visit and at the end of the study.

Signs and symptoms of adverse events were closely monitored during treatment cycles. Safety laboratory measures were done at Screening, during the 72hr hospitalization (first cycle), at every interim visit , and at the end of the study. A follow-up safety visit was to be scheduled at least 30 days after the end of treatment.

CAP-232 plasma levels were also determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV kidney clear cell carcinoma.
* Confirmed progressive disease after receiving a previous systemic therapy, including at least one line of standard of care.
* Measurable disease
* Age >18 years.
* Life expectancy of greater than 3 months.
* At least 5 years free of any other cancer(s). Basal cell carcinoma, provided that is neither infiltrating nor sclerosing and carcinoma in situ of the cervix, is acceptable.
* ECOG performance status 2 or lower (Karnofsky 60%).
* Normal organ and marrow function
* Adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and have the willingness to sign a written informed consent document.
* Ability to receive central vein access catheter and manage an infusion pump.
* Women of child bearing potential must have a negative serum pregnancy test.

Exclusion Criteria:

* Anti-cancer therapy within 4 weeks prior to entering the study
* Investigational agents less than 30 days prior to enrollment in the study.
* Known brain metastases
* History of allergic reactions attributed to compounds of similar composition to CAP-232.
* Past or current cancer other than kidney cancer, except for: Curatively treated non-melanoma skin cancer, In situ carcinoma of the cervix, Other cancer curatively treated and with no evidence of disease for at least 5 years
* Uncontrolled intercurrent illness /social situations that would limit compliance with study requirements.
* Breastfeeding
* Patients previously enrolled into this study and subsequently withdrawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter was the response rate based on RECIST criteria after 3 cycles

SECONDARY OUTCOMES:
Safety (through clinical and biological evaluations)
Other efficacy parameters (progression-free survival rate, time to progression and overall survival)
Pharmacokinetic (PK) characteristics of the first 15 recruited patients
Quality of life
Biological modulation (through potential blood and/or urine biomarkers including M2PK)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Guillot, MD, Principal Investigator — Institut de Cancérologie de la Loire, Dpt Oncologie Médicale, Saint-Priest en Jarez, France; Damien Pouessel, MD, Principal Investigator — CRLC Val d'Aurelle Paul-Lamarque, Montpellier, France
Locations (2):
- France (2):
  - CRLC Val d'Aurelle Paul-Lamarque, Montpellier
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Tejeda M, Gaal D, Hullan L, Hegymegi-Barakonyi B, Keri G. Evaluation of the antitumor efficacy of the somatostatin structural derivative TT-232 on different tumor models. Anticancer Res. 2006 Sep-Oct;26(5A):3477-83. PMID 17094470
- [Background] Tejeda M, Gaal D, Hullan L, Csuka O, Schwab R, Szokoloczi O, Keri G. A comparison of the tumor growth inhibitory effect of intermittent and continuous administration of the somatostatin structural derivative TT-232 in various human tumor models. Anticancer Res. 2006 Jul-Aug;26(4B):3011-5. PMID 16886628
- [Background] Gyergyay F, Gödény M, Sármay G, Kralovanszky J, Papp E, Gergye M, Vincze B, Kéri G, Bodrogi I : Antitumor activity and pharmacology of TT-232 (a novel somatostatin structural derivative) in malignant melanoma patients JCO, 2004 ASCO Annual Meeting Proceedings Vol 22, No 14S (July 15 Supplement), 2004: 3151